CLINICAL TRIAL: NCT01281007
Title: A Prospective, Randomized, Multicenter Study of the Efficacy and Safety of Famciclovir 125 mg Comparing to Aciclovir 200 mg in Patients With Active Recurrent Genital Herpes
Brief Title: Efficacy of Oral Famciclovir 125mg Comparing to Aciclovir 200 mg Treatment in Patients With Active Recurrent Genital Herpes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F125EMS1010
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Results first posted 2015-07-07 (Estimated); Last update posted 2021-04-21 (Actual); Status verified 2015-07

CONDITIONS: GENITAL HERPES
Keywords: Herpes Simplex Virus
MeSH Terms: conditions — Herpes Genitalis; Herpes Simplex | interventions — Famciclovir; Acyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Famciclovir 125 mg (Experimental): 1 tablet every 12 hours for 5 days
  Interventions: Drug: Famciclovir
- Aciclovir 200 mg (Active Comparator): 1 tablet every 4 hours (excluding nocturnal dose) for 5 days
  Interventions: Drug: Aciclovir

INTERVENTIONS:
Drug: Famciclovir — Famciclovir 125 mg every 12 hours for 5 days
  Arms: Famciclovir 125 mg
Drug: Aciclovir — Aciclovir 200 mg every 4 hours fo 5 days
  Arms: Aciclovir 200 mg

SUMMARY:
Recurrent genital herpes is a commonly occurring sexually transmitted disease caused by herpes simplex virus (HSV). There are effective oral prescription antiviral medicines available to reduce the discomfort of symptoms, such as famciclovir and aciclovir.

This is a phase III, multicenter, randomized, parallel-group study to compare the efficacy and safety of treatment with famciclovir (125 mg) versus aciclovir (200 mg) in patients with active recurrent genital herpes.

DETAILED DESCRIPTION:
STUDY DESIGN

* Open-label, prospective, parallel group, intent to treat trial
* Experiment duration: 5 days
* 2 visits (days 1, and 5)
* Reduction of symptoms
* Adverse events evaluation

ELIGIBILITY:
Inclusion criteria:

1. Patients must be able to understand the study procedures agree to participate and give written consent.
2. Patients with clinical diagnosis of recurrent genital herpes;
3. Score symptoms higher than 4;
4. Negative pregnant urine test.

Exclusion criteria:

1. Pregnancy or risk of pregnancy.
2. Lactation
3. Any pathology or past medical condition that can interfere with this protocol.
4. Non-steroidal anti-inflammatory drug , hormonal anti-inflammatory or immunosuppressive drugs (in the last 30 days and during the study);
5. Patients with immunodeficiency and/or immunosuppressive disease;
6. Hypersensitivity to components of the formula;
7. Other conditions deemed reasonable by the medical investigator as to the disqualification of the individual from study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-07; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Amazonas, MD, Study Director — EMS
Locations (9):
- Brazil (9):
  - Centro de Medicina Reprodutiva Dr Carlos Isaia Filho Ltda, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - SPVita, Bragança Paulista, São Paulo
  - Caep Centro Avancado de Estudos E Pesquisas Ltda, Campinas, São Paulo
  - CEMICAMP - Centro de Pesquisas em Saúde Reprodutiva de Campinas, Campinas, São Paulo
  - CECIP - Centro de Estudos Clínicos do Interior Paulista, Jaú, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirao Preto da Universidade de Sao Paulo, Ribeirão Preto, São Paulo
  - Instituto Sirio Libanes de Ensino e Pesquisa, São Paulo, São Paulo
  - Afip - Associacao Fundo de Incentivo A Psicofarmacologia, São Paulo, São Paulo

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Famciclovir 125 mg | Aciclovir 200 mg
Started | 75 | 75
Completed | 71 | 67
Not Completed | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Famciclovir 125 mg | Aciclovir 200 mg | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 73 | 143
  >=65 years | 5 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 50 | 107
  Male | 18 | 25 | 43
Region of Enrollment [Number; unit: participants]
  Brazil | 75 | 75 | 150

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Will be Evaluated by the Proportion of Subjects With Non Herpes Manifestation
Description: Symptoms evaluated: erythema, papule, vesicle, ulcer, crust, or healed skin.
Time Frame: Day 5
Measure: Number; unit: subjects
Arm/Group | Famciclovir 125 mg | Aciclovir 200 mg
Number analyzed (Participants) | 75 | 75
subjects | 73 | 52

2. Secondary Outcome: Safety Will be Evaluated by the Adverse Events Occurence
Description: Adverse events will be collected and followed in order to evaluate safety and tolerability
Time Frame: Day 5
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Famciclovir 125 mg | Aciclovir 200 mg
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 10/75 | 12/75
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Famciclovir 125 mg (N=75) | Aciclovir 200 mg (N=75)
Headache (Nervous system disorders) | 10 (10) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No